CLINICAL TRIAL: NCT06131918
Title: Assessment of Resveratrol, Alpha Lipoic Acid and Superoxide Dismutase on Oxidative Stress Biomarkers in Type 2 Diabetes Mellitus Patients With Neuropathy: A Randomized Control Trial
Brief Title: Assessment of Antioxidant Therapy on Oxidative Stress Biomarkers in Type 2 Diabetic Patients With Neuropathy
Acronym: RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAMIDHABIB
Record Dates: First submitted 2023-08-25; First posted 2023-11-14 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Diabetic Neuropathy
Keywords: Diabetic Neuropathy; Resveratrol; Alpha lipoic acid; Superoxide dismutase
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Resveratrol; Thioctic Acid; Superoxide Dismutase

STUDY DESIGN:
Intervention Model Description: Four parallel treatment arms will be included.
Who Masked: Participant
Masking Description: The participants will not be given information about the medication.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resveratrol+ Alpha lipoic acid +Superoxide dismutase (Active Comparator): This group will receive Resveratrol 1500 mg BD Tab Alpha lipoic acid 600 mg BD Tab Superoxide dismutase 250 mg BD
  Interventions: Drug: Resveratrol, Alpha lipoic acid, Super oxide dismutase
- Resveratrol (Active Comparator): This group will receive Tab Resveratrol 1500 mg BD
  Interventions: Drug: Resveratrol
- Alpha lipoic Acid (Active Comparator): This group will receive Tab Alpha lipoic acid 600mg BD
  Interventions: Drug: Alpha lipoic acid
- Superoxide dismutase (Active Comparator): This group will receive Tab Superoxide dismutase 250mg BD
  Interventions: Drug: Super Oxide Dismutase

INTERVENTIONS:
Drug: Resveratrol, Alpha lipoic acid, Super oxide dismutase — Tab Resveratrol 1500 mg BD Tab Alpha lipoic Acid 600 mg BD Tab Superoxide dismutase 250 mg BD
  Other Names: Resveratrol; Alpha lipoic Acid; Superoxide dismutase
  Arms: Resveratrol+ Alpha lipoic acid +Superoxide dismutase
Drug: Resveratrol — Tab Resveratrol 1500 mg BD Tab Placebo 600mg BD Cap Placebo 250mg BD
  Other Names: Tab Resveratrol; Tab Placebo; Capsule Placebo
  Arms: Resveratrol
Drug: Alpha lipoic acid — Tab Alpha lipoic acid 600 mg BD Tab Placebo 600mg BD Cap Placebo 250mg BD
  Other Names: Tab Placebo; Cap Placebo
  Arms: Alpha lipoic Acid
Drug: Super Oxide Dismutase — Tab Super oxide dismutase 250 mg BD Tab Placebo 600mg BD Cap Placebo 250mg BD
  Other Names: Superoxide dismutase; Tab Placebo; Cap Placebo
  Arms: Superoxide dismutase

SUMMARY:
Type 2 DM subjects having numbness, tingling and paresthesia in hands and feet (neuropathy) will be recruited. Screening of neuropathy will be done by Michigan screening instrument. This will be followed by nerve conduction studies. Specific blood parameters will also be checked. The subjects will then be divided into four treatment arms. Three groups will receive single drug and the fourth one will receive all the three drugs. These will be given for four months. Follow up will be done every month. At the end of four months, they will be assessed for any improvement in neuropathy by using Michigan neuropathy instrument and nerve conduction studies. Blood parameters will also be measured again.

DETAILED DESCRIPTION:
Type 2 DM subjects having numbness, tingling and paresthesia in hands and feet (neuropathy) will be recruited. They will be screened by Michigan neuropathy scale. This is tool used for screening neuropathy. Subjects having a score equal to or greater then 4 will be examined for further evaluation. This will be followed by nerve conduction studies for objective assessment of neuropathy. For inclusion criteria the test performed will be HbA1c, CBC, ESR, RFTs and LFTs. After screening the baseline levels of Superoxide radical, Super oxide dismutase, Glutathione peroxidase and Malonaldehyde will be measured. The subjects will be randomly divided into four treatment arms. Group A will receive Triple regime antioxidant therapy including Resveratrol 1500 mg two times a day, Alpha lipoic acid 600 mg two times a day and Superoxide dismutase 250 mg once a day. Group B will receive Resveratrol 1500mg BD, Group C will be on Tab Alpha lipoic acid 600 mg BD and Group D will take Superoxide dismutase once a day. The subjects will be kept blinded about the medication. They will be followed every month in which their quality of life will be assessed using Nottingham health profile and neuropathy will be assessed by Michigan neuropathy scale. At the end of four months blood tests will again be performed to check the levels of Superoxide radical, Superoxide dismutase, Glutathione peroxidase and Malonaldehyde. NCS will be done to see any improvement in neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus
* Age between 40-60 years

Exclusion Criteria:

* Malignancy
* Vitamin B12 deficiency
* History of drug or alcohol abuse
* Taking antioxidant treatment
* History and baseline investigations for renal hepatic and haematological diseases
* Pregnant or lactating women.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Change in nerve conduction latency, velocity and amplitude. | 4 months
  This will be assessed by doing Nerve conduction studies at the start and end of trial. The nerves examined will be Median and Ulnar nerves in upper limb both for motor and sensory conduction. In case of lower limbs motor nerve Peroneal and sensory Sural nerve will be examined.
Change in clinical symptoms of neuropathy. | 4 months
  1. It will be assessed by Michigan neuropathy screening instrument at the start of the trial, at the end of each month and at the conclusion of the trial.
  2. Changes in Quality of life will be assessed by Nottingham health profile.
  3. Safety and tolerability of treatment. Recording and evaluation of adverse events and side effects will be done throughout the treatment period

SECONDARY OUTCOMES:
levels of superoxide radical anion, | 4 months
  Change in the levels of superoxide radical anion
Levels of Malonaldehyde oxidative stress biomarker | 4 months
  Change in the levels of oxidative stress biomarkers
Levels of Superoxide dismutase and Glutathione peroxidase | 4 months
  Change in the levels of antioxidant enzymes

CONTACTS AND LOCATIONS:
Overall Officials: Syed Hamid Habib, PhD, Study Director — Khyber Medical University
Locations (1):
- Syed Hamid Habib, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang B, Guo L, Li BY, Zhen JH, Song J, Peng T, Yang XD, Hu Z, Gao HQ. Resveratrol attenuates early diabetic nephropathy by down-regulating glutathione s-transferases Mu in diabetic rats. J Med Food. 2013 Jun;16(6):481-6. doi: 10.1089/jmf.2012.2686. PMID 23767859
- [Background] Bhatt JK, Thomas S, Nanjan MJ. Resveratrol supplementation improves glycemic control in type 2 diabetes mellitus. Nutr Res. 2012 Jul;32(7):537-41. doi: 10.1016/j.nutres.2012.06.003. Epub 2012 Jul 27. PMID 22901562
- [Background] Kennedy DO, Wightman EL, Reay JL, Lietz G, Okello EJ, Wilde A, Haskell CF. Effects of resveratrol on cerebral blood flow variables and cognitive performance in humans: a double-blind, placebo-controlled, crossover investigation. Am J Clin Nutr. 2010 Jun;91(6):1590-7. doi: 10.3945/ajcn.2009.28641. Epub 2010 Mar 31. PMID 20357044
- [Background] Szkudelski T, Szkudelska K. Resveratrol and diabetes: from animal to human studies. Biochim Biophys Acta. 2015 Jun;1852(6):1145-54. doi: 10.1016/j.bbadis.2014.10.013. Epub 2014 Oct 27. PMID 25445538
- [Background] Bjornholm M, Zierath JR. Insulin signal transduction in human skeletal muscle: identifying the defects in Type II diabetes. Biochem Soc Trans. 2005 Apr;33(Pt 2):354-7. doi: 10.1042/BST0330354. PMID 15787605
- [Background] Villegas-Rivera G, Roman-Pintos LM, Cardona-Munoz EG, Arias-Carvajal O, Rodriguez-Carrizalez AD, Troyo-Sanroman R, Pacheco-Moises FP, Moreno-Ulloa A, Miranda-Diaz AG. Effects of Ezetimibe/Simvastatin and Rosuvastatin on Oxidative Stress in Diabetic Neuropathy: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Oxid Med Cell Longev. 2015;2015:756294. doi: 10.1155/2015/756294. Epub 2015 Jul 28. PMID 26290682
- [Background] Oyenihi AB, Ayeleso AO, Mukwevho E, Masola B. Antioxidant strategies in the management of diabetic neuropathy. Biomed Res Int. 2015;2015:515042. doi: 10.1155/2015/515042. Epub 2015 Mar 2. PMID 25821809
- [Background] Kumar A, Kaundal RK, Iyer S, Sharma SS. Effects of resveratrol on nerve functions, oxidative stress and DNA fragmentation in experimental diabetic neuropathy. Life Sci. 2007 Mar 6;80(13):1236-44. doi: 10.1016/j.lfs.2006.12.036. Epub 2007 Jan 20. PMID 17289084
- [Background] Xiao WH, Bennett GJ. Effects of mitochondrial poisons on the neuropathic pain produced by the chemotherapeutic agents, paclitaxel and oxaliplatin. Pain. 2012 Mar;153(3):704-709. doi: 10.1016/j.pain.2011.12.011. Epub 2012 Jan 13. PMID 22244441
- [Background] Pham-Huy LA, He H, Pham-Huy C. Free radicals, antioxidants in disease and health. Int J Biomed Sci. 2008 Jun;4(2):89-96. PMID 23675073
- [Background] Valko M, Leibfritz D, Moncol J, Cronin MT, Mazur M, Telser J. Free radicals and antioxidants in normal physiological functions and human disease. Int J Biochem Cell Biol. 2007;39(1):44-84. doi: 10.1016/j.biocel.2006.07.001. Epub 2006 Aug 4. PMID 16978905
- [Background] Rahimi-Madiseh M, Malekpour-Tehrani A, Bahmani M, Rafieian-Kopaei M. The research and development on the antioxidants in prevention of diabetic complications. Asian Pac J Trop Med. 2016 Sep;9(9):825-831. doi: 10.1016/j.apjtm.2016.07.001. Epub 2016 Aug 5. PMID 27633293